CLINICAL TRIAL: NCT05384613
Title: Evaluation of Quality Indicators on Analgesia, Sedation and Delirium in Intensive Care Patients and Their Impact on Outcome Indicators and Economic Indicators
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: ECOPAD
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Delirium; Pain
Keywords: Sedation
MeSH Terms: conditions — Delirium; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective cohort study to investigate the adherence to the process indicators for pain management, sedation management and management of delirium on outcome indicators and cost/revenues in individual patients and subcohorts.

DETAILED DESCRIPTION:
The evaluation of quality-related process indicators (in this case, Quality Indicator II of the Intensive Care Quality Indicators of the DIVI*: Management of Analgesia, Sedation and Delirium) will be correlated with economic parameters of the treatment from economic data (DRG revenue, case costs). Data from clinical routine care from the Charite hospital systems will be used with further analysis of outcome indicators from routine data (e.g. 30-day readmission rate, mortality, infection rate, length of stay). The aim of the study is to identify and evaluate incentive mechanisms for the implementation of quality-relevant care processes using the example of adherence to a quality indicator regarding management of analgesia, sedation and delirium) on detailed cost shares and case proceeds. In addition, further routine data, which may represent influencing factors like comorbidities (Charlson Comorbitity Index) are calculated using the ICD-10 coding. Also procedures using the OPS system are evaluated.

In this retrospective cohort study, patient records from the clinical information systems from 2012 to 2021 will be analyzed.. The analysis is also intended to analyze whether alternatively, cross-treatment outcome indicators can be defined, which would demonstrate not only positive patient-oriented results but also positive economic results as a potential incentive for health care service providers.

(* DIVI: Deutsche Interdisziplinäre Vereinigung für Intensiv- und Notfallmedizin = German Interdisciplinary Association for Intensive Care and Emergency Medicine)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Exclusion Criteria:

* Incomplete electronic records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Electronically documented anesthesiological or intensive care treatment in the HIS (Hospital Information System) and PDMS (Patient Data Management System) of the Charité (Dep. for Anesthesiology with focus on operative intensive care, CCM/CVK) from 01.01.2012- 31.12.2021
Sampling Method: Probability Sample
Enrollment: 20220 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Influence of compliance to a quality indicator (Monitoring sedation, analgesia, delirium) | 01.01.2012- 31.12.2021
  Influence of compliance to a quality indicator (Quality Indicator II of the DIVI; Management of Analgesia, Sedation and Delirium) and the relationship to case specific revenues and case costs according to case-specific analysis based on hospital financial data

SECONDARY OUTCOMES:
Comorbidity scores | 01.01.2012- 31.12.2021
  (Comorbidity scores are assessed according to Charlson comorbidity index (CCI) employing routine data, like icd-10 codes.
Outcome indicators | 01.01.2012- 31.12.2021
  Outcome indicators from routine data are e. g. 30-day readmission rate, mortality, infection rate, length of stay, etc. )

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zuber A, Rubarth K, Forster F, Balzer F, Spies C, Furstenau D, Kumpf O. The impact of adhering to a quality indicator for sedation, analgesia, and delirium management on costs, revenues, and clinical outcomes in intensive care in Germany: A retrospective observational study. PLoS One. 2024 Aug 15;19(8):e0308948. doi: 10.1371/journal.pone.0308948. eCollection 2024. PMID 39146321